CLINICAL TRIAL: NCT02623998
Title: An Open-label, Randomized, Parallel Design Trial to Compare the Efficacy of a Sitagliptin-based Metabolic Intervention Versus Standard Diabetes Therapy in Inducing Remission of Type 2 Diabetes
Brief Title: Remission Evaluation of a Metabolic Intervention in Type 2 Diabetes With Sitagliptin (REMIT-Sita)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMIT-Sita
Record Dates: First submitted 2015-12-04; First posted 2015-12-08 (Estimated); Results first posted 2022-03-14 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Insulin; Glargine; Metformin; Sitagliptin; Diet; Excercise; Lifestyle
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Insulin Glargine; Sitagliptin Phosphate; Metformin; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination; Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Drug: insulin glargine - sc injection Drug: sitagliptin/metformin - oral administration Behavioral: lifestyle therapy
  Interventions: Drug: insulin glargine; Drug: sitagliptin/metformin; Behavioral: lifestyle therapy
- Standard Care (No Intervention): Standard glycemic care as informed by the current clinical practice guidelines

INTERVENTIONS:
Drug: insulin glargine — Dose is titrated to achieve fasting normoglycemia
  Other Names: Lantus
  Arms: Intervention
Drug: sitagliptin/metformin — Dose is titrated to 50/1000 mg bid or maximal tolerated dose
  Other Names: Janumet
  Arms: Intervention
Behavioral: lifestyle therapy — Lifestyle intervention includes individualized dietary and exercise advice and frequent visits for goal reinforcement, behavior modification and problem-solving
  Other Names: diet and exercise
  Arms: Intervention

SUMMARY:
The purpose of the study is to determine whether in patients with early type 2 diabetes,a short-term intensive metabolic intervention comprising of sitagliptin, metformin, basal insulin glargine and lifestyle approaches will be superior to standard diabetes therapy in achieving sustained diabetes remission.

DETAILED DESCRIPTION:
This is a multicentre, open-label, randomized controlled trial in 100 patients with recently-diagnosed T2DM. Participants will be randomized to 2 treatment groups: (a) a 12-week course of treatment with sitagliptin, metformin, insulin glargine and lifestyle therapy, or (b) standard diabetes therapy, and followed for a total of 64 weeks (1 year and 3 months). In all participants with HbA1C < 7.3% at the 12 week visit, glucose-lowering medications will be discontinued and participants will be encouraged to continue with lifestyle modifications and regular glucose monitoring. Participants with HbA1C ≥ 7.3% at this visit or who meet criteria for hyperglycemic relapse after stopping drugs will receive standard glycemic management as informed by the current Canadian Diabetes Association clinical practice guidelines

ELIGIBILITY:
Inclusion Criteria:

1. men and women 30-80 years of age inclusive;
2. type 2 diabetes mellitus diagnosed by a physician within 5 years prior to patient enrollment;
3. anti-diabetic drug regimen (either drug or dose of drug) unchanged during 8 weeks prior to screening and randomization;
4. HbA1C ≤ 9.5% on no oral hypoglycemic agents or HbA1C ≤ 8.0% on 1 oral agent or on half-maximal doses of 2 agents;
5. body mass index ≥ 23 kg/m2;
6. a negative pregnancy test and an agreement to use a reliable method of birth control for the duration of the trial in all females with childbearing potential;
7. ability and willingness to perform self-monitoring of capillary blood glucose (SMBG); ability and willingness to self-inject insulin;
8. provision of informed consent.

Exclusion Criteria:

1. current use of insulin;
2. history of hypoglycemia unawareness; history of severe hypoglycemia requiring assistance within the last 5 years;
3. renal dysfunction as evidenced by serum creatinine (Cr) ≥ 124 μmol/l;
4. history of lactic acidosis or diabetic ketoacidosis;
5. active liver disease or elevated alanine transferase (ALT) levels ≥ 2.5 times upper limit of normal at the time of enrollment;
6. history of pancreatitis;
7. cardiovascular disease including any of: a) systolic blood pressure > 180 mmHg or diastolic blood pressure > 105 mmHg; b) peripheral vascular disease; c) left bundle branch block or second or third degree AV block; d) tachyarrhythmias or bradyarrhythmias with uncontrolled ventricular rate; e) stenotic valvular heart disease; f) cardiomyopathy; g) history of heart failure; h) history of aortic dissection; i) documented history of angina or coronary artery disease; j) history of stroke or transient ischemic attack;
8. history of any disease requiring continuous systemic glucocorticoid treatment;
9. history of any major illness with a life expectancy of < 3 years;
10. history of injury or any other condition that significantly limits participant's ability to achieve moderate levels of physical activity;
11. excessive alcohol consumption (>14 alcoholic drinks per week in men and >7 alcoholic drinks per week in women);
12. known hypersensitivity to insulin glargine, metformin, or any DPP-4 inhibitor.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-07-09 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia McInnes, MD, Principal Investigator — McMaster University; Hertzel C Gerstein, MD, Study Chair — Hamilton Health Sciences Corporation
Locations (6):
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - Health Science Centre, Winnipeg, Manitoba
  - McMaster University, Hamilton, Ontario
  - St. Joseph's Hospital, London, Ontario
  - LMC, Markham, Ontario
  - Univeristy of Montreal, Montreal, Quebec

REFERENCES:
- [Derived] McInnes N, Hall S, Hramiak I, Sigal RJ, Goldenberg R, Gupta N, Rabasa-Lhoret R, Braga M, Woo V, Sultan F, Otto R, Smith A, Sherifali D, Liu YY, Gerstein HC; REMIT-sita Collaborative Group. Remission of Type 2 Diabetes Following a Short-term Intensive Intervention With Insulin Glargine, Sitagliptin, and Metformin: Results of an Open-label Randomized Parallel-Design Trial. Diabetes Care. 2022 Jan 1;45(1):178-185. doi: 10.2337/dc21-0278. PMID 34728531

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Standard Care
Started | 50 | 52
Completed | 48 | 51
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Standard Care | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (8.7) | 54.7 (9.3) | 55.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 32 | 32 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 42 | 47 | 89
  Non-Caucasian | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  Canada | 50 | 52 | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hyperglycemia Relapse in the Experimental Group Compared to the Control Group
Description: Hyperglycemia relapse for primary outcome was defined as any one of:
  1. Capillary glucose >10 mmol/L on >/=50% of readings over 1 week;
  2. HbA1C >/=6.5%;
  3. use of diabetes drugs;
  4. fasting plasma glucose >/= 7.0 mmol/L;
  5. 2-hour postprandial plasma glucose >/=11.1 mmol/L on an oral glucose tolerance test.
Time Frame: 64 weeks of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 50 | 52
Participants | 41 | 48

2. Primary Outcome: Number of Participants With Severe Hypoglycemic Episodes
Time Frame: 64 weeks of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 50 | 52
Participants | 0 | 0

3. Secondary Outcome: Number of Participants Achieving Drug-free Diabetes Remission
Description: Diabetes remission is defined as absence of hyperglycemia relapse
Time Frame: 24 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 50 | 52
Participants | 8 | 4

4. Secondary Outcome: Number of Participants With Drug-free Normal Glucose Tolerance
Description: Normal glucose tolerance is defined as a FPG<6.1 mmol/L and a 2-hour plasma glucose <7.8 mmol/L on a 75 g oral glucose tolerance test
Time Frame: 24 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 50 | 52
Participants | 3 | 1

5. Secondary Outcome: Percent Change in Weight
Time Frame: Baseline and 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 50 | 52
% change | -2.1 (2.5) | -1.4 (2.9)

6. Secondary Outcome: Change in Waist Circumference
Time Frame: Baseline and 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 50 | 52
cm | -2.3 (3.5) | -1.8 (4.8)

ADVERSE EVENTS:
Time Frame: 64 weeks
Arm/Group | Intervention | Standard Care
All-Cause Mortality (participants affected / at risk) | 1/50 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/52
Other Adverse Events (participants affected / at risk) | 9/50 | 4/52
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=50) | Standard Care (N=52)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Anxiety/depression (Psychiatric disorders) | 1 (1) | 1 (1)
Vasovagal syncope (Cardiac disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (2)
Allergic conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Elective surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Superficial skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-12-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT02623998/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT02623998/SAP_001.pdf